CLINICAL TRIAL: NCT03510078
Title: Intensive Versus Conventional Hyperglycemic Control in Hospitalized Non-critically Ill Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Irit Ayalon Dangur, MD, Dr, Internal Medicine Doctor, Principal Investigator, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0695-17-RMC
Record Dates: First submitted 2018-03-25; First posted 2018-04-27 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Diabetes Mellitus; Non-critically Ill Patients
Keywords: Diabetes Mellitus; hyperglycemic control; hospitalization; internal medicine
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive glycemic control (Experimental): With a target of blood glucose range of 130 mg/dL or less
  Interventions: Drug: Insulin
- Conventional glycemic control (Experimental): With a target of blood glucose range of 130-180 mg/dL
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Insulin — Insulin for glycemic control according to the allocation

SUMMARY:
Hyperglycemia is a common condition among hospitalized patients. The occurrence of severe hyperglycemia is associated with increased morbidity and mortality in several populations. Several trials assessed the benefits of aggressive versus conventional glucose control. These studies evaluated different patient populations, glucose targets and treatment protocols and as a result reported conflicting results. To date there are no clear guidelines regarding to the preferred glucose target range in hospitalized non-critically ill patients. The common practice is to maintain glucose level lower than 180 mg/dl however there are no evidence based regarding to the outcomes of hospitalized patients treated with intensive compared to conventional glycemic control. This prospective randomized controlled study will compare intensive vs. standard glycemic control in hospitalized non-critically ill patients.

Within 24 hours of hospitalization in the internal medical or geriatric departments, patients who are expected to require hospitalization for at least three consecutive days will be randomly assigned into one of the two study groups - intensive with a target blood glucose range of 130 mg per deciliter or less, or conventional glucose control, with a target of 130-180 mg per deciliter. The investigators defined the primary end point as a composite outcome of mortality in 30 days, severe hypoglycemia, severe infections within 30 days, CVA and cardiac ischemic events within 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18 years old.
* History of type 2 diabetes mellitus for at least three months or a blood glucose level of 200 mg per deciliter or higher in two different consecutive measurements.
* A minimum of three days of hospitalization.

Exclusion Criteria:

* Diabetic ketoacidosis or hyperosmolar non-ketotic state at any stage of hospitalization.
* Patients expected to require intensive care unit admission or immediate surgical intervention.
* History of current drug or alcohol abuse.
* History of current mental illness.
* Child-bearing potential or a positive urine pregnancy test.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2018-04-17 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Composite outcome of: 1. mortality in 30 days | 30 days
Severe hypoglycemia | 30 days
Severe infections | 30 days
  Severe infections will be defined as a hospitalization as a result of sepsis, pneumonia or soft tissue infection or other infection requiring intravenous antibiotic therapy that occurred during hospitalization.
Cerebro-Vascular accidents | 30 days
Cardiac ischemic events | 30 days

SECONDARY OUTCOMES:
Each component of the primary outcomes | 30 days
Repeat hospitalizations within 90 days | 90 days
  Repeated hospitalizations will be defined as the number of repeated hospitalizations in 90 days.
Severe infections within 90 days | 90 days
  Severe infections will be defined as a hospitalization as a result of sepsis, pneumonia or soft tissue infection or other infection requiring intravenous antibiotic therapy that occurred during hospitalization.
Length of hospitalization | 90 days
  Will be measured as the number of days from the admission to the discharge from hospital.

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Rambam Medical Center, Haifa
  - Rabin Medical Center, Petah Tikva

IPD SHARING:
Plan to Share IPD: No